CLINICAL TRIAL: NCT02229864
Title: ABSORB III RCT Pharmacokinetics (PK) Sub-study
Brief Title: Pharmacokinetics of Everolimus in Absorb BVS in Patients With Coronary Artery Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-392 B
Record Dates: First submitted 2014-06-09; First posted 2014-09-03 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis; Coronary Disease; Coronary Stenosis
Keywords: Absorb™ BVS; Angioplasty; Bioabsorbable; BVS; Coronary Artery Disease; Coronary Artery Endothelial Responsiveness; Coronary artery restenosis; Coronary artery stenosis; Coronary scaffold; Coronary Stent; Drug eluting stents; Everolimus; Myocardial ischemia; Stent thrombosis; Stents
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Disease; Coronary Restenosis; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Coronary artery stenting: Absorb BVS (Experimental): Subjects receiving Absorb Bioresorbable Vascular Scaffold (BVS)
  Interventions: Device: Coronary artery stenting: Absorb BVS

INTERVENTIONS:
Device: Coronary artery stenting: Absorb BVS — * Scaffold diameters: 2.5, 3.0 and 3.5 mm
  * Scaffold lengths: 8, 12, 18, and 28 mm

SUMMARY:
The ABSORB III PK sub-study is a prospective, open-label, non-blinded study enrolling approximately 12 subjects in up to 5 US sites. ABSORB III PK sub-study is a part of ABSORB III RCT (NCT01751906). The objective is to determine the pharmacokinetics of everolimus delivered by the Absorb BVS in a separate and non-randomized cohort of subjects who only receive Absorb BVS with a maximum of two de novo native coronary artery lesions after implantation of the Absorb BVS.

Note: The ABSORB III PK subjects will not contribute to the determination of the ABSORB III RCT primary endpoint.

DETAILED DESCRIPTION:
To ensure the PK measurements reflect everolimus exposure due to Absorb BVS only, the PK sub-study will not allow non-target lesion treatment.

Blood Sampling Timing:

* Pre-Absorb BVS implantation: Baseline

  o Baseline is defined as prior to implantation of the first Absorb BVS; the blood sample will be drawn on the day of the index procedure either through a heparin lock, venous sheath, or venipuncture.
* Post-Absorb BVS implantation: 10 and 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 24 hrs (1 day), 48 hrs (2 days), 72 hrs (3 days), 96 hrs (4 days), 120 hrs (5 days), 168 hrs (7 days), 336 hrs (14 days), and 720 hrs (30 days).

  * Post-implantation blood samples will be drawn at the time intervals stated above; timing of the post-implantation sampling will begin when the last Absorb BVS is deployed, i.e. last Absorb BVS delivery catheter is removed from the body.

Pharmacokinetic (PK) parameters will include time to maximum concentration (tmax); maximum concentration (Cmax); AUC24h: Area under the blood analyte concentration vs. time curve from time 0 up to 24 hours post placement of the last Absorb BVS; AUClast: Area under the blood analyte concentration vs. time curve from time 0 up to the last quantifiable concentration; AUC 0-infinity: Area under the blood analyte concentration vs. time curve from time zero and extrapolated to infinite time; terminal elimination rate constant (λz); terminal elimination half-life (t1/2term); drug clearance (CL).

ELIGIBILITY:
General Inclusion Criteria:

1. 18 years of age.
2. Subject or a legally authorized representative must provide written Informed Consent prior to any study related procedure, per site requirements.
3. Evidence of myocardial. In the absence of noninvasive ischemia, FFR must be done and indicative of ischemia.
4. An acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Female subject of childbearing potential who does not plan pregnancy for up to 1 year following the index procedure.
6. Female subject is not breast-feeding at the time of the screening visit and will not be breast-feeding for up to 1 year following the index procedure.
7. Subject agrees to not participate in any other investigational or invasive clinical study for a period of 1 year following the index procedure.

Angiographic Inclusion Criteria:

1. One or two de novo target lesions:

   1. If two target lesions are present, they must be present in different epicardial vessels and both must satisfy the angiographic eligibility criteria.
   2. The definition of epicardial vessels means the left anterior descending (LAD), left coronary artery (LCX), and right coronary artery (RCA) and their branches. Thus, the patient must not have lesions requiring treatment in e.g. both the LAD and a diagonal branch.
2. Target lesion(s) must be located in a native coronary artery with a visually estimated or quantitatively assessed % diameter stenosis (DS) of ≥ 50% and < 100% with a thrombolysis in myocardial infarction (TIMI) flow of ≥ 1 and one of the following: stenosis ≥ 70%, an abnormal functional test (e.g., fractional flow reserve (FFR), stress test), unstable angina or post-infarct angina.

   1. Lesion(s) must be located in a native coronary artery with reference vessel diameter (RVD) by visual estimation of ≥ 2.50 mm and ≤ 3.75 mm.
   2. Lesion(s) must be located in a native coronary artery with length by visual estimation of ≤ 24 mm.

General Exclusion Criteria:

1. Any surgery requiring general anesthesia or discontinuation of aspirin and/or an Adenosine diphosphate receptor (ADP) antagonist is planned within 12 months after the procedure.
2. Subject has known hypersensitivity or contraindication to device material and its degradants (everolimus, poly (L-lactide), poly (DL-lactide), lactide, lactic acid) and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated. Subject has a known contrast sensitivity that cannot be adequately pre-medicated.
3. Subject has known allergic reaction, hypersensitivity or contraindication to aspirin; or to clopidogrel and prasugrel and ticagrelor; or to heparin and bivalirudin, and therefore cannot be adequately treated with study medications.
4. Subject had an acute myocardial infarction (AMI: STEMI or NSTEMI) within 72 hours of the index procedure and both creatine kinase (CK) and creatine kinase myocardial-band isoenzyme (CK-MB) have not returned to within normal limits at the time of index procedure; or subject with stable angina or silent ischemia has CK-MB that is greater than normal limits at the time of the index procedure.
5. Subject is currently experiencing clinical symptoms consistent with new onset AMI (STEMI or NSTEMI), such as nitrate-unresponsive prolonged chest pain with ischemic ECG changes.
6. Subject has a cardiac arrhythmia as identified at the time of screening for which at least one of the following criteria is met:

   1. Subject requires coumadin or any other agent for chronic oral anticoagulation
   2. Subject is likely to become hemodynamically unstable due to their arrhythmia
   3. Subject has poor survival prognosis due to their arrhythmia
7. Subject has a left ventricular ejection fraction (LVEF) < 30%
8. Subject has undergone prior percutaneous coronary intervention (PCI) within the target vessel(s) during the last 12 months.
9. Subject requires future staged PCI either in target or non-target vessels or subject requires future peripheral interventions < 30 days after the index procedure.
10. Subject has received any solid organ transplants or is on a waiting list for any solid organ transplants.
11. At the time of screening, the subject has a malignancy that is not in remission.
12. Subject is receiving immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.). Note: corticosteroids are not included as immunosuppressant therapy.
13. Subject has previously received or is scheduled to receive radiotherapy to a coronary artery (vascular brachytherapy), or the chest/mediastinum.
14. Subject is receiving or will require chronic anticoagulation therapy (e.g., coumadin, dabigatran, apixaban, rivaroxaban or any other agent for any reason).
15. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3.
16. Subject has a documented or suspected hepatic disorder as defined as cirrhosis or Child-Pugh ≥ Class B.
17. Subject has renal insufficiency as defined as an estimated glomerular filtration rate (GFR) < 30 ml/min/1.73m2 or dialysis at the time of screening.
18. Subject is high risk of bleeding for any reason; has a history of bleeding diathesis or coagulopathy; has had a significant gastro-intestinal or significant urinary bleed within the past six months.
19. Subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past six months, or any prior intracranial bleed, or any permanent neurologic defect, or any known intracranial pathology (e.g., aneurysm, arteriovenous malformation, etc.).
20. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion. Note: femoral arterial disease does not exclude the patient if radial access may be used.
21. Subject has life expectancy < 5 years for any non-cardiac cause or cardiac cause.
22. Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason.
23. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
24. Subject is part of a vulnerable population

Angiographic Exclusion Criteria:

All exclusion criteria apply to the target lesion(s) or target vessel(s).

1. Lesion which prevents successful balloon pre-dilatation
2. Lesion is located in left main.
3. Aorto-ostial RCA lesion.
4. Lesion located within 3 mm of the origin of the LAD or LCX.
5. Lesion involving a bifurcation with a:

   1. side branch ≥ 2 mm in diameter, or
   2. side branch with either an ostial or non-ostial lesion with diameter stenosis > 50%, or
   3. side branch requiring dilatation.
6. Anatomy proximal to or within the lesion that may impair delivery of the Absorb BVS.
7. Vessel contains thrombus as indicated in the angiographic images or by intravascular ultrasound (IVUS) or optical coherence tomography (OCT).
8. Lesion or vessel involves a myocardial bridge.
9. Vessel has been previously treated with a stent at any time prior to the index procedure such that the Absorb BVS would need to cross the stent to reach the target lesion.
10. Vessel has been previously treated and the target lesion is within 5 mm proximal or distal to a previously treated lesion.
11. Target lesion located within an arterial or saphenous vein graft or distal to any arterial or saphenous vein graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G. Rizik, MD, Principal Investigator — Scottsdale Healthcare, Scottsdale, AZ; Louis A. Cannon, MD, Principal Investigator — Cardiac and Vascular Research Center of Northern Michigan Petoskey, MI
Locations (2):
- United States (2):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on June 2, 2014 and the last subject was enrolled on September 17, 2014. The last 30-day follow-up visit occurred on October 14, 2014. Database was locked on Oct 29, 2014.
Pre-assignment Details: In this sub-study, subjects received either one (N=8) or two (N=4) Absorb BVS with the diameters of 2.5, 3.0 and 3.5 mm and lengths of 8, 12, 18 and 28 mm. The total everolimus dose ranged from 181 μg to 443 μg.
Groups:
- Coronary Artery Stenting: Absorb BVS: Subjects receiving Absorb Bioresorbable Vascular Scaffold (BVS)
  Coronary artery stenting: Absorb BVS: • Scaffold diameters: 2.5, 3.0 and 3.5 mm
  • Scaffold lengths: 8, 12, 18, and 28 mm
Period: Overall Study
Arm/Group | Coronary Artery Stenting: Absorb BVS
Started | 12
Completed | 9
Not Completed | 3
Not completed — Death | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The PK sub-study had slightly more male subjects, and slightly more subjects with dyslipidemia and hypertension requiring medication and subjects with stable angina as compared to ABSORB III Primary Analysis Group. The PK sub-study had fewer subjects who had undergone prior coronary intervention.
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Hypertension Requiring Medication [Count of Participants; unit: Participants] | 12
Dyslipidemia Requiring Medication [Count of Participants; unit: Participants] | 12
Prior Coronary Intervention [Count of Participants; unit: Participants] | 1
Stable Angina [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax)
Description: Maximal observed blood analyte concentration. Cmax is the highest blood everolimus concentration reached during the 30 day period of the study after assessing at different time frames (10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, and 30 days post implantation).
Time Frame: 0 to 30 days
Population: ITT population. The number of participants analyzed includes subjects who had available follow-up data at that time frame.
Measure: Median (Full Range); unit: nanograms per milliliter
Groups:
- Coronary Artery Stenting: Absorb BVS: Subjects receiving Absorb Bioresorbable Vascular Scaffold (BVS).
  Absorb BVS with the diameters of 2.5, 3.0 and 3.5 mm and lengths of 8, 12, 18 and 28 mm. The total everolimus dose ranged from 181 μg to 443 μg.
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
nanograms per milliliter | 2.397 [1.085 to 4.460]

2. Primary Outcome: Time of Maximum (Tmax)
Description: Time to reach the maximal observed blood analyte concentration during the 30 day period of the study after assessing at different time frames (10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, and 30 days post implantation).
Time Frame: 0 to 30 days
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
Hours | 0.55 [0.17 to 2.37]

3. Primary Outcome: AUC24h
Description: Area under the blood analyte concentration vs. time curve from time 0 up to 24 hours post placement of the last Absorb BVS. Calculated by the Lin Up Log Down trapezoidal method.
Time Frame: 0 to 24 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
ng*h/mL | 22.67 [12.09 to 44.22]

4. Primary Outcome: AUC Last
Description: Area under the blood analyte concentration vs. time curve from time 0 up to the last quantifiable concentration reached during the 30 day period of the study. After assessing at different time frames (10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, and 30 days post implantation). Calculated by the Lin Up Log Down trapezoidal method.
Time Frame: 0 to 30 days
Population: as for outcome 1
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
ng*h/mL | 55.90 [25.37 to 104.6]

5. Primary Outcome: AUC 0-infinity
Description: AUC 0-infinity: Area under the blood analyte concentration vs. time curve from time zero and extrapolated to infinite time, reached during the 30 day period of the study. After assessing at different time frames (10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, and 30 days post implantation).
  calculated as: AUC0-∞ = AUClast + (Clast/λz)
  The percentage of AUC0-∞ obtained by extrapolation (%AUC0-∞ex) is calculated as:
  %AUC0-∞ex = (AUC0-∞ - AUClast)/ AUC0-∞ * 100
Time Frame: 0 to 30 days
Population: as for outcome 1
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
ng*h/mL | 72.02 [33.15 to 120.8]

6. Primary Outcome: Terminal Elimination Rate Constant (λz)
Description: The apparent terminal elimination rate constant during the 30 day period of the study. After assessing at different time frames (10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, and 30 days post implantation). Determined by linear regression of terminal points of the ln-linear analyte concentration-time curve.
Time Frame: 0 to 30 days
Population: as for outcome 1
Measure: Median (Full Range); unit: 1/hour
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
1/hour | 0.01092 [0.006027 to 0.01511]

7. Primary Outcome: Terminal Elimination Half-life (t1/2term)
Description: The apparent terminal elimination half-life, reached during the 30 day period of the study. After assessing at different time frames (10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, and 30 days post implantation).
  calculated as: t1/2term = 0.693/λz.
Time Frame: 0 to 30 days
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
Hours | 63.5 [45.9 to 115.0]

8. Primary Outcome: Drug Clearance (CL)
Description: The systemic drug clearance, reached during the 30 day period of the study. After assessing at different time frames (10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, and 30 days post implantation).
  Calculated as: CL = Dose/AUC0 - ∞ .
Time Frame: 0 to 30 days
Population: as for outcome 1
Measure: Median (Full Range); unit: Liter/hour
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
Liter/hour | 3.451 [2.421 to 5.460]

9. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Target Lesion Failure (TLF) includes Cardiac Death, Target vessel - myocardial infarction and Target Lesion Revascularization (TLR).
Time Frame: 0 to 1853 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 11
Participants | 2

10. Secondary Outcome: Number of Participants With All Death
Description: All death includes cardiac death, vascular death, and non-cardiac death.
Time Frame: 0 to 1853 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 11
Participants | 2

11. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI)
Description: All myocardial infarction includes target vessel myocardial infarction (TV-MI) and not attributable to target vessel myocardial infarction (NTV-MI).
Time Frame: 0 to 1853 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 11
Participants | 4

12. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: All target lesion revascularization includes ischemia-driven target lesion revascularization (ID-TLR) and non ischemia-driven target lesion revascularization (NID-TLR).
Time Frame: 0 to 1853 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 11
Participants | 0

13. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: All target vessel revascularization includes ischemia driven target vessel revascularization (ID-TVR) and non ischemia driven target vessel revascularization (NID-TVR).
Time Frame: 0 to 1853 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 11
Participants | 1

14. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization includes ischemia driven revascularization and non ischemia driven revascularization.
Time Frame: 0 to 1853 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 11
Participants | 3

15. Secondary Outcome: Number of Participants With Acute Stent/Scaffold Thrombosis (Definite/Probable)
Description: Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Acute scaffold/stent thrombosis : 0 - 24 hours post stent implantation Subacute scaffold/stent thrombosis: >24 hours - 30 days post stent implantation Late scaffold/stent thrombosis: 30 days - 1 year post stent implantation Very late scaffold/stent thrombosis: >1 year post stent implantation
Time Frame: ≤ 1 day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
Participants | 0

16. Secondary Outcome: Number of Participants With Subacute Stent/Scaffold Thrombosis (Definite/Probable)
Description: as for outcome 15
Time Frame: >1 to 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
Participants | 0

17. Secondary Outcome: Number of Participants With Late Stent/Scaffold Thrombosis (Definite/Probable)
Description: as for outcome 15
Time Frame: 31 to 393 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 12
Participants | 0

18. Secondary Outcome: Number of Participants With Cumulative Stent/Scaffold Thrombosis (Definite/Probable)
Description: as for outcome 15
Time Frame: 0 to 1853 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Stenting: Absorb BVS
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Coronary Artery Stenting: Absorb BVS
All-Cause Mortality (participants affected / at risk) | 2/12
Serious Adverse Events (participants affected / at risk) | 10/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coronary Artery Stenting: Absorb BVS (N=12)
ANGINA PECTORIS (Cardiac disorders) | 1
ANGINA PECTORIS AGGRAVATED (Cardiac disorders) | 1
ARRHYTHMIA (Cardiac disorders) | 1
ATRIAL FIBRILLATION AGGRAVATED (Cardiac disorders) | 1
ATRIAL FIBRILLATION WITH RAPID VENTRICULAR RESPONSE (Cardiac disorders) | 1
NON STEMI (Cardiac disorders) | 1
STABLE ANGINA PECTORIS (Cardiac disorders) | 1
UNSTABLE ANGINA (Cardiac disorders) | 1
SMALL BOWEL OBSTRUCTION (Gastrointestinal disorders) | 1
UPPER GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1
CHEST PAIN (General disorders) | 1
CHEST PAIN (NON-CARDIAC) (General disorders) | 1
BRONCHITIS (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
CELLULITIS OF LEG (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 3
PAINFULL ARM (Musculoskeletal and connective tissue disorders) | 1
SPINAL STENOSIS OF LUMBAR REGION (Musculoskeletal and connective tissue disorders) | 1
ACUTE ON CHRONIC RENAL FAILURE (Renal and urinary disorders) | 1
ACUTE RENAL FAILURE (Renal and urinary disorders) | 1
BENIGN PROSTATIC HYPERTROPHY (Reproductive system and breast disorders) | 1
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1
POPLITEAL VEIN THROMBOSIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coronary Artery Stenting: Absorb BVS (N=12)
ANGINA PECTORIS (Cardiac disorders) | 3
ANGINA PECTORIS AGGRAVATED (Cardiac disorders) | 1
ARRHYTHMIA (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
ATRIAL FIBRILLATION AGGRAVATED (Cardiac disorders) | 1
ATRIAL FIBRILLATION WITH RAPID VENTRICULAR RESPONSE (Cardiac disorders) | 1
BRADYCARDIA (Cardiac disorders) | 1
CHEST PAIN - CARDIAC (Cardiac disorders) | 2
CONGESTIVE HEART FAILURE (Cardiac disorders) | 1
CORONARY ARTERY DISSECTION (Cardiac disorders) | 3
CORONARY NO-REFLOW PHENOMENON (Cardiac disorders) | 1
NON STEMI (Cardiac disorders) | 1
STABLE ANGINA PECTORIS (Cardiac disorders) | 1
UNSTABLE ANGINA (Cardiac disorders) | 1
HEARTBURN (Gastrointestinal disorders) | 1
SMALL BOWEL OBSTRUCTION (Gastrointestinal disorders) | 1
TOOTHACHE (Gastrointestinal disorders) | 1
UPPER GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1
CHEST PAIN (General disorders) | 1
CHEST PAIN (NON-CARDIAC) (General disorders) | 4
INFUSION SITE HEMATOMA (General disorders) | 1
BRONCHITIS (Infections and infestations) | 2
CELLULITIS (Infections and infestations) | 1
CELLULITIS OF LEG (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
BRUISE (Injury, poisoning and procedural complications) | 1
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 1
POSTOPERATIVE HYPOTENSION (Injury, poisoning and procedural complications) | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1
TICK BITE (Injury, poisoning and procedural complications) | 1
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1
CARDIAC ENZYMES INCREASED (Investigations) | 2
CREATINE KINASE MB INCREASED (Investigations) | 3
BACK PAIN AGGRAVATED (Musculoskeletal and connective tissue disorders) | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 3
MONOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
PAINFUL L ARM (Musculoskeletal and connective tissue disorders) | 1
SPINAL STENOSIS OF LUMBAR REGION (Musculoskeletal and connective tissue disorders) | 1
DIZZINESS (Nervous system disorders) | 1
SCIATICA (Nervous system disorders) | 1
ACUTE ON CHRONIC RENAL FAILURE (Renal and urinary disorders) | 1
ACUTE RENAL FAILURE (Renal and urinary disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
BENIGN PROSTATIC HYPERTROPHY (Reproductive system and breast disorders) | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
OBSTRUCTIVE SLEEP APNEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1
HYPOTENSION (Vascular disorders) | 1
POPLITEAL VEIN THROMBOSIS (Vascular disorders) | 1
SLOW REFLOW PHENOMENON (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators shall not present or publish, nor submit for publication, any work resulting from the Services without Sponsor's prior written approval.

Except as specifically set forth herein, neither party shall use the other party's name or trademark, or the name nor trademark of such other party's affiliate, in any publicity, advertising or announcement, or disclose the existence or terms of this Agreement, without the consenting party's prior written approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT02229864/Prot_SAP_000.pdf